CLINICAL TRIAL: NCT06022172
Title: The Effect of Motivational Interviewing Based on the Calgary Family Intervention Model on Care Burden, Self-Efficacy and Coping With Stress in Parents of Children With Cerebral Palsy
Brief Title: Calgary Model Motivational Interviewing for Parents of Children With CP Care Burden Self-efficacy Coping With Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Igdir University (Other)
Collaborators: Kafkas University (Other)
Responsible Party: Principal Investigator, Gülçin Aşut, Teaching Assistant, Igdir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gulcin1
Record Dates: First submitted 2023-08-14; First posted 2023-09-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy
Keywords: SP Ebeveyn Calgary Model Bakım Verme Öz-Yeterlik Stres
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 30 people in the experimental group and 30 people in the control group, a total of 60 people will be included in the study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): MOTIVATIONAL INTERVIEW BASED ON THE CALGARY FAMILY INTERVENTION MODEL IN PARENTS WITH A CHILD WITH CEREBRAL PALS.
  Interventions: Diagnostic Test: MOTIVATIONAL INTERVIEW BASED ON THE CALGARY FAMILY INTERVENTION MODEL IN PARENTS WITH A CHILD WITH CEREBRAL PALS.
- CONTROL GROUP (No Intervention): no action will be taken

INTERVENTIONS:
Diagnostic Test: MOTIVATIONAL INTERVIEW BASED ON THE CALGARY FAMILY INTERVENTION MODEL IN PARENTS WITH A CHILD WITH CEREBRAL PALS. — Motivational interview based on Calgary family intervention model in parents of children with cerebral palsy.
  Introductory information form, caregiving burden, parent self-efficacy and stress coping styles scale will be used.
  Arms: Experimental group

SUMMARY:
Cerebral palsy (CP) is a non-progressive problem that occurs as a result of damage or lesion in the brain tissue in the prenatal, perinatal or postnatal periods for any reason, causing permanent impairment in the development of posture and movement. In addition to the impairments in the motor area in CP; It can be seen in problems such as perception, cognitive, sensory, communication, social, behavioral, musculoskeletal, epilepsy .Parents who are primary caregivers of the child with CP; They have a very important caregiver role in meeting the processes such as the treatment of the child, daily life needs and rehabilitation.Parental self-efficacy has been defined as the judgments and beliefs held by the parents to cope with the difficulties they experience in raising and caring for children with developmental disabilities and to reach the goal.The long process of caring for the child with cerebral palsy and the dependence of the child on the parent increase the stress of the caregivers. The Calgary Family Intervention Model (CAMM), one of the nursing models, is the first family intervention model in the field of nursing. The model focuses on improving, developing and maintaining the family's functionality in three areas. These three areas are cognitive, emotional and behavioral.

DETAILED DESCRIPTION:
Cerebral palsy is a problem that causes permanent impairment in the development of non-progressive posture and movement, which occurs as a result of damage or lesion in the brain tissue for any reason in prenatal, perinatal or postnatal periods. In addition to the disorders in the motor area in SP; It can be seen in problems such as perception, cognitive, sensory, communication, social, behavioral, musculoskeletal, epilepsy .

Parents who are primary caregivers of the child with CP; They have a very important caregiver role in meeting the processes such as the treatment of the child, daily life needs and rehabilitation . Meeting all these special needs of the child with CP creates the burden of care for the parents .

Parental self-efficacy has been defined as the judgments and beliefs held by the parents to cope with the difficulties they experience in raising and caring for children with developmental disabilities and to reach the goal . People with high parental self-efficacy; It has been stated that they are more self-confident in taking and fulfilling their parenting duties, they make more effort, and they focus more on a solution in the face of any problem. The long process of caring for the child with cerebral palsy and the dependence of the child on the parent increase the stress of the caregivers. Caregiving stress affects the physiological, psychological, economic and social behaviors of parents.

The Calgary Family Intervention Model, one of the nursing models, is the first family intervention model in the field of nursing. The model focuses on improving, developing and maintaining the family's functionality in three areas. These three areas are cognitive, emotional and behavioral. The Calgary Family Intervention Model is an important model in increasing family functionality and providing change in pediatric nursing practice .

In the literature review, no other study has been found yet, examining the effect of motivational interviewing based on the Calgary Family Intervention model on the burden of care, self-efficacy and coping with stress in parents of children with cerebral palsy. It is believed that the motivational interview technique to be applied to the parents can be more beneficial for the children they care for and themselves, by revealing the effects of the disease, the responsibilities brought by the disease, the care burden arising from these responsibilities, parent self-efficacy and coping with stress.

Materials and Methods This study is a randomized controlled study. The research will be carried out in the interview rooms of the rehabilitation centers with the parents of children with cerebral palsy whose children attend a special rehabilitation center in the province of Iğdır.

The universe of the research will be the parents of 120 children with cerebral palsy between the ages of 6-18 who attend private rehabilitation centers in the province of Iğdır. Without using any sample selection method in the research, parents who meet the inclusion criteria and participate voluntarily in the research will be considered as the sample of the research. The number of samples was calculated in G*Power program. There is no similar research in the related literature. As a result of the power analysis performed before the study, the number of people to be included in the study group for percentage 80 power was calculated as 26. At least 30 parents will be included in both groups for possible sample loss during the implementation phase of the research. A list will be created by assigning a code number to each parent.

Personal information form, caregiving burden scale, Parental Self-Efficacy Scale, and Ways of Coping with Stress Scale developed by the researchers will be used to collect research data.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with cerebral palsy between the ages of 6-18,
* Able to read and write Turkish, accessible and able to communicate,
* Orientation and cooperation
* Hearing, comprehension and vision problems,
* Parents who agreed to participate in the study were determined as .

Exclusion Criteria:

* Having difficulty in communication
* Not being literate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pre-test data collection | Time frame 1 or 2 months.
  The research pre-test data will be carried out by the researcher between September 2023 and October 2023 in the interview rooms of rehabilitation centers, with the parents of children with cerebral palsy attending a private rehabilitation center in Iğdır. Introductory information form The burden of care for individuals in the experimental and control groups in data collection, parent self-efficacy scale and coping styles scale will be applied. In the care burden scale, a minimum score of 0 and a maximum of 88 points can be obtained from the scale. The lowest score in the self-efficacy scale is 17 and the highest score is 119. In the scale of coping with stress, the total score is calculated is not done.
Collection of post-test data | Time frame one or two months.
  The motivational interview based on the Calgary family intervention model for each parent in the experimental group will consist of 6 sessions lasting 45 minutes, one week apart. After the interviews, the final test will be held after the last session and 15 days later. Parents of children with cerebral palsy whose children attend a special rehabilitation center in Istanbul will meet in the meeting rooms of the rehabilitation centers. Introductory information form, caregiver burden scale, parent self-efficacy scale and coping styles scale will be used to collect data.
  A score of 88 can be obtained. The lowest score in the self-efficacy scale is 17, and the highest score is 119. The total score is not calculated in the scale of coping with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Aşut, Doctorate, Principal Investigator — Igdir University
Locations (1):
- Igdir university, Iğdır, Turkey (Türkiye)